CLINICAL TRIAL: NCT02424786
Title: Non-adherence and Polypharmacy in Elderly Patients With Chronic Renal Failure: Predictors and an Intervention
Brief Title: Non-adherence and Polypharmacy in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Krystina Parker, MD, pHD-student, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-068
Record Dates: First submitted 2015-03-31; First posted 2015-04-23 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Adherence
Keywords: Adherence; Polypharmacy; Elderly; Chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Potentially Inappropriate Medication List

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Other): Medication lists from the patients randomized in the intervention group will be evaluated by the research physician with the help of STOPP/START criteria.
  Feedback of this screening will be given to the team responsible for patient treatment.
  Interventions: Other: STOPP/START criteria
- Control (No Intervention): Patients in this arm will receive standard pharmacological treatment

INTERVENTIONS:
Other: STOPP/START criteria — Evaluation of medication lists
  Arms: Intervention group

SUMMARY:
The study aims to investigate adherence and polypharmacy in elderly patients with chronic kidney disease (CKD) and End Stage Renal Disease (ESRD). The investigators look into possible factors or predictors that may affect adherence and reduce polypharmacy. Factors could be: quality of life, anxiety and depression, beliefs about medicine and cognitive impairment.

The investigators are planning an intervention with the screening tool Screening Tool of Older Person's potentially inappropriate Prescription/Screening tool to Alert to Right Treatment (STOPP/START ) criteria to evaluate medication lists of the participating patients.

DETAILED DESCRIPTION:
The investigators intend to include all patients > 65 years old, in dialysis treatment (hemodialysis and peritoneal dialysis), as well as patients with CKD stage 5.

The recruitment will be done as follows:

The patients will be screened according to inclusion criteria. Afterwards each patient will be invited to a first meeting that explains the aim of the study, giving the opportunity for discussion and consideration, and presenting the consent information. After giving the consent the patient will be invited to a second meeting with blood tests, data registration, medication registration, undergoing MMS and handing over the questionnaires forms.

Randomization:

After the initial assessment and compliance with the eligibility criteria, participants will be randomized into an intervention group (medication list will be evaluated by STOPP/START criteria) and a control group (medication list will not be evaluated by STOPP/START criteria). Randomization numbers will be generated by a random number generator. A series of numbered, sealed, opaque envelopes will be used to ensure confidentiality. Each envelope will contain a card with information about the group allocation. The group allocation is concealed from the researcher and patients at baseline registration.

Each patients will get questionnaires for: Quality of life using Kidney Disease Quality of Life - Short form 36 (KDQOL-Short form 36 ) and EuroQoL-3D (EQ-3D), beliefs about medicine, Hospital Anxiety and Depression Scale (HADS), Morisky medication adherence scale and visual adherence scale (VAS), sleeping related questionnaires (Epworth, Berlin, Pittsburgh). A Mini Mental Status (MMS) test will be done regarding cognitive function.

Each patients will get the opportunity to have a polysomnograph for one night.

With STOPP/START criteria the medication list will be evaluated for the patients who are randomized in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* All patients > 65 years with CKD, stage 5 (eGFR ≤ 12 ml/min), or undergoing treatment with hemodialysis and peritoneal dialysis

Exclusion Criteria:

* Patients not willing to participate
* Patients diagnosed with dementia or severe cognitive disorder (MMS < 25),
* Patients with hearing impairment
* Patients with language difficulties

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-05; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Prevalence for medication non-adherence | 6 months - 1 year
  Adherence measured by Morisky medication adherence scale and visual adherence scale

SECONDARY OUTCOMES:
Improvement of polypharmacy | 1-2 year
  Randomization of all patients into intervention group and control group. Comparing both groups by using STOPP/START criteria with the aim to assess numbers of patients with inappropriate medications
Improvement of adherence | 1-2 year
  Randomization of all patients into intervention group and control group with the aim to improve adherence by using Morisky medication adherence scale and visual adherence scale
Association between beliefs about medication and anxiety and depression with medication non-adherence and quality of life | 1-2 years
  Questionnaires about: Beliefs about medicine, depression and anxiety (measured by HADS), quality of life (measured by KDQOL-Short form 36, EQ-5D), and adherence (measured by Morisky medication adherence scale and visual adherence scale)
Predictors for medication non-adherence | 6 months - 1 year
  Questionnaires about depression and anxiety (HADS)
Risk factors for medication non-adherence | 6 months - 1 year
  Questionnaires about beliefs about medicine
Medication non-adherence risk factors | 6 months - 1 year
  Questionnaires about sleep quality (Epworth, Berlin, Pittsburgh questionnaires)
Non-adherence and medication - predictors | 6 months - 1 year
  Questionnaires about quality of life measured by KDQOL-Short form 36 and EQ-5D

OTHER OUTCOMES:
Change from baseline regarding prescription of inappropriate medications in the intervention group | baseline and 6 months
  Improvement of polypharmacy
Change from baseline in Morisky medication adherence scale and visual adherence scale | baseline
  Difference between Morisky medication scale score and score from the Visual adherence score

CONTACTS AND LOCATIONS:
Overall Officials: Knut Stavem, Professor, Principal Investigator — University Hospital, Akershus; Ingrid Os, Principal Investigator — Univeristy Hospital, Ullevål
Locations (3):
- Norway (3):
  - Vestre Viken Sykehus, Drammen
  - University Hospital, Ullevål, Oslo
  - University Hospital, Akershus, Oslo

IPD SHARING:
Plan to Share IPD: No
No data will be shared

REFERENCES:
- [Derived] Parker K, Bull-Engelstad I, Benth JS, Aasebo W, von der Lippe N, Reier-Nilsen M, Os I, Stavem K. Effectiveness of using STOPP/START criteria to identify potentially inappropriate medication in people aged >/= 65 years with chronic kidney disease: a randomized clinical trial. Eur J Clin Pharmacol. 2019 Nov;75(11):1503-1511. doi: 10.1007/s00228-019-02727-9. Epub 2019 Jul 29. PMID 31359099